CLINICAL TRIAL: NCT04346602
Title: A Study on the Clinical and Psychological Characteristics of Patients With COVID-2019
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Doctor, Jilin University
Other Study IDs: 130004
Record Dates: First submitted 2020-04-06; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-2019
Keywords: COVID-2019; clinical; psychological; symptom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with COVID-2019: Patients with COVID-2019 would be observed.
  Interventions: Other: all treatment about COVID-2019

INTERVENTIONS:
Other: all treatment about COVID-2019 — All patients with COVID-2019 would receive treatment provided by the government and should comply with relevant laws and regulations.

SUMMARY:
A study on the clinical and psychological characteristics of patients with coronavirus disease 2019 (COVID-2019)

DETAILED DESCRIPTION:
The main objective of this study is to study the clinical and psychological responses of patients with COVID-2019 during the whole treatment process. Including clinical symptoms, auxiliary examination results, and corresponding psychological changes, including depression, anxiety, insomnia, etc. This study will draw lessons about treatment and other better advices for other countries and regions.

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID-2019

Exclusion Criteria:

* No

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with COVID-2019 would be observed.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
fever | one month
  The fever is one main clinical characteristics of patients with COVID-2019, Measured by thermometer. 37.2-38 degrees Celsius, low fever; 38-39 degrees Celsius, moderate fever; 39-40 degrees Celsius, high fever.

SECONDARY OUTCOMES:
cough | one month
  Cough is one main symptom of patients with COVID-2019. "Yes" or "no" would be recorded.
diarrhea | one month
  Diarrhea is one symptom of some patients with COVID-2019. "Yes" or "no" would be recorded.
anxiety | two months
  Anxiety is one main psychological characteristic of patients with COVID-2019. It would be assessed by Hamilton anxiety scale (HAMA). Scores of HAMA were positively correlated with the severity of anxiety.
insomnia | two months
  Insomnia is one main psychological characteristic of patients with COVID-2019. It would be assessed by Athens insomnia scale (AIS). Scores of AIS were positively correlated with the severity of insomnia.
depression | two months
  Depression is one psychological characteristic of patients with COVID-2019.It would be assessed by Hamilton Depression Rating Scale (HAMD) . Scores of HAMD were positively correlated with the severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Yang, Master, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan B, Song L, Guo J, Wang Y, Peng L, Li D. Association Between Clinical Characteristics and Short-Term Outcomes in Adult Male COVID-19 Patients With Mild Clinical Symptoms: A Single-Center Observational Study. Front Med (Lausanne). 2021 Jan 5;7:571396. doi: 10.3389/fmed.2020.571396. eCollection 2020. PMID 33469542